CLINICAL TRIAL: NCT04867746
Title: HamRepair: Clinical and Functional Outcomes at Least 2 Years After Hamstring Muscle Repair
Brief Title: Clinical and Functional Outcomes at Least 2 Years After Hamstring Muscle Repair
Acronym: HamRepair
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02276; mu21Stoffel2
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Hamstring Muscle Repair; Hamstring Rupture
Keywords: postoperative muscular imbalances; muscular deficits; pathological gait; Isokinetic muscle strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection by health questionnaires — Health questionnaires to assess scores concerning pain and function of the treated leg and overall health
Other: assessment of muscle strength — Muscle strength will be measured bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA). For the knee, maximum isokinetic flexion and extension torques will be collected between full extension and full flexion at a movement speed of 60°/s (5 repetitions) and 240°/s (15 repetitions). Maximum joint torques in each movement direction will be recorded for each joint and normalized to body weight.
Other: assessment of gait — Instrumented gait analysis on a treadmill with an embedded plantar pressure plate (h/p/cosmos, Zebris FDM-T, Isny, Germany; 7168 sensors; area, 1.5 * 0.5 m; range, 1-120 N/cm2; precision, 1-120 N/cm2 ± 5%; sampling rate, 120 Hz) and on an overground walkway with two embedded force plates (Kistler force plate 9260AA6, Kistler AG, Winterthur, Switzerland; sampling rate 2400 Hz). Simultaneously with the plantar pressure or force data, kinematic and electromyographic (EMG) data will be collected. Participants will then walk for 1 minute at their preferred walking speed (0% slope and at 15% slope) and at 1.2 m/s (0% slope). For all conditions, kinematic, EMG and pressure data will be recorded for 1 minute. Subsequently, the treadmill speed will be increased to preferred running speed and 2.3 m/s (0% slope), and data for 1 minute running will be recorded. Subjects will then complete overground walking and running trials on the walkway with embedded force plates.
Other: assessment of squatting and single leg hops — Participants perform three jumps on a force plate. Maximum jump length, Maximum flexion and extension angles and joint moments will be identified. Subsequently, participants perform three squats onto two force plates (one per foot). On- and off times will be computed for each muscle and condition.
Other: assessment of postural stability — The length of the centre of pressure path will be measured during two 30-second unipedal stance trials using a force plate.

SUMMARY:
This study is to evaluate functional outcomes of a new, intraoperative lateral positioning of the anchors on the tuber ischiadicum, in comparison to regular anatomical anchoring direct on top of the tuber ischiadicumafter hamstring muscle repair. This study is to quantify at least 2 years postoperative functional, biomechanical and clinical outcomes including side-to-side differences in muscle strength, unipedal balance, gait, jumping and squatting function, muscle activity, in patients treated by hamstring muscle repair.

DETAILED DESCRIPTION:
The design of this pilot study is a descriptive cross-sectional single centre analysis involving all patients previously treated with hamstring repair. All of these patients will be asked to participate in clinical and detailed functional analysis at least 2 years after surgery. Specifically, biomechanical and functional data including isokinetic muscle strength, clinical scores, ROM, joint kinematics and kinetics during walking, running, squatting and single leg jumps, muscle activity and single leg balance ability in the affected and contralateral leg will be collected. These parameters will be compared between legs and correlated with clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years since hamstring muscle repair

Exclusion Criteria:

* Revision surgery within 6 months before testing on the ipsilateral knee and hip
* BMI > 35 kg/m2
* Previous injury and surgical procedures of the contralateral knee and hip within the last year
* Neuromuscular disorders affecting lower limb movement
* Additional pathologies that influence the mobility of the lower extremity
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated between 11/2014 and 04/2019 (n=17) with hamstring muscle repair at the Department of Orthopaedics and Traumatology, University Hospital Basel will be contacted at least 2 years after surgery by the treating surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength | at baseline (total timeframe for each participant approx 150 minutes)
  Isokinetic muscle strength deficit of the knee flexors and extensors in the injured leg compared to the contralateral leg, assessed by a dynamometer

SECONDARY OUTCOMES:
Range of motion of the knee (degree) | at baseline (total timeframe for each participant approx 150 minutes)
  Range of motion of the knee in comparison to the contralateral leg
Range of motion of the hip (degree) | at baseline (total timeframe for each participant approx 150 minutes)
  Range of motion of the hip in comparison to the contralateral leg
Joint kinematics (maximum flexion and extension angles) | at baseline (total timeframe for each participant approx 150 minutes)
  Joint kinematics (in walking and running) in comparison to the contralateral leg
Muscle activity (intensity of the electromyographic signals) | at baseline (total timeframe for each participant approx 150 minutes)
  Muscle activity (in gait, balance, squatting and single leg hopping) in comparison to the contralateral leg

OTHER OUTCOMES:
Perth Hamstring Assessment Tool | at baseline (total timeframe for each participant approx 20 minutes)
  The Perth Hamstring Assessment Tool (PHAT) is to evaluate functional outcomes of proximal hamstring re-attachment surgery. The PHAT provides a score out of 100, with a higher score corresponding to higher function. The questionnaire uses a visual analogue scale for pain scores as well as categorical scores for activity levels.
EQ-5D-5L | at baseline (total timeframe for each participant approx 20 minutes)
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Lower Extremity Functional Scale (LEFS) | at baseline (total timeframe for each participant approx 20 minutes)
  The Lower Extremity Functional Scale (LEFS) is intended to assess functional status in patients with disability of the lower extremity. It is a 20 item questionnaire. The maximum score obtainable is 80 which means complete function and the lowest score is 0 which means very low and severely impaired function.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stoffel, Prof. Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Mauch M, Nuesch C, Buhl L, Chocholac T, Mundermann A, Stoffel K. Reconstruction of proximal hamstring ruptures restores joint biomechanics during various walking conditions. Hip Int. 2024 Jul;34(4):516-523. doi: 10.1177/11207000241230282. Epub 2024 Feb 19. PMID 38372148
- [Derived] Chocholac T, Buhl L, Nuesch C, Bleichner N, Mundermann A, Stoffel K. Modified surgical anchor refixation in older patients with acute proximal hamstring rupture: clinical outcome, patient satisfaction and muscle strength. Arch Orthop Trauma Surg. 2023 Aug;143(8):4679-4688. doi: 10.1007/s00402-022-04752-3. Epub 2023 Jan 9. PMID 36622424